CLINICAL TRIAL: NCT02565836
Title: Reversal of Warfarin-associated Major Hemorrhage: a Multicenter, Retrospective Cohort Study of Fixed-dose Activated (FEIBA VH) Versus Variable-dose Inactivated (Kcentra) Prothrombin Complex Concentrate
Brief Title: Fixed-dose Activated Versus Variable-dose Inactivated Prothrombin Complex Concentrate for Warfarin-associated Major Bleed
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 15092404
Record Dates: First submitted 2015-09-24; First posted 2015-10-01 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Hemorrhage
Keywords: Vitamin K 1; prothrombin complex concentrates; warfarin
MeSH Terms: conditions — Hemorrhage | interventions — anti-inhibitor coagulant complex

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- fixed-dose aPCC: Patients receiving fixed-dose activated prothrombin complex concentrate (FEIBA VH) for reversal of warfarin-associated major hemorrhage.
  Interventions: Drug: fixed-dose activated prothrombin complex concentrate
- variable-dose PCC: Patients receiving vairable-dose inactivated prothrombin complex concentrate (Kcentra) for reversal of warfarin-associated major hemorrhage.
  Interventions: Drug: variable-dose inactivated prothrombin complex concentrate

INTERVENTIONS:
Drug: fixed-dose activated prothrombin complex concentrate — FEIBA VH 500 units IV one time for INR less than 5. FEIBA VH 1000 units IV one time for INR greater than 5.
  Check INR after infusion and may repeat dose if INR still elevated
  Other Names: FEIBA; FEIBA VH
  Groups: fixed-dose aPCC
Drug: variable-dose inactivated prothrombin complex concentrate — Kcentra 25 units/kg IV one time for INR less than 4. Kcentra 35 units/kg IV one-time for INR 4 to 6. Kcentra 50 units/kg IV one-time for INR greater than 6.
  Check INR after infusion and may repeat dose if INR still elevated.
  Other Names: Kcentra
  Groups: variable-dose PCC

SUMMARY:
This study aims to assess a fixed-dose regimen of activated prothrombin complex concentrate (FEIBA VH, Baxter) versus the variable, manufacturer recommended, dose regimen of inactivated prothrombin complex concentrate (Kcentra, CSL Behring) for reversal of warfarin-associated major hemorrhage.

DETAILED DESCRIPTION:
Warfarin, a vitamin K antagonist (VKA), is the most frequently prescribed oral anticoagulant. Warfarin-associated major hemorrhage occurs at a rate of 1.7% to 3.4% in routine clinical practice and warrants rapid reversal of anticoagulation by correcting supratherapeutic international normalized ratio (INR) values.

Warfarin inhibits synthesis of vitamin K dependent coagulation factors II, VII, IX, and X, and strategies for reversal of warfarin-associated coagulopathy are aimed at restoring deficient factors. Four-factor prothrombin complex concentrates (PCCs) contain the coagulation factors which warfarin inhibits and are an attractive option for rapid reversal due to ease of reconstitution and no requirement for blood-type matching.

Manufacturer dosing recommendations exist for PCCs based on patient weight, baseline INR, and target INR, but studies have suggested fixed dosing strategies in an effort to determine the most efficacious dose for VKA-reversal while sparing adverse events. These studies have also utilized different PCC formulations, with some studies utilizing 4-factor activated PCC (aPCC), which denotes product containment of factor VII in an activated state.

In the United States, product availability is limited to a single 4-factor aPCC (FEIBA VH, Baxter) indicated for hemophilia patients with inhibitors and a single 4-factor inactivated PCC (Kcentra, CSL Behring) approved for VKA-reversal. Various institutions choose to utilize off-label fixed dosing strategies of 4-factor aPCC in an effort to administer the lowest possible dose to reverse VKAs, while others utilize manufacturer recommended dosing of 4-factor inactivated PCC.

ELIGIBILITY:
Inclusion Criteria:

* Pre-treatment INR lab value greater than 1.5
* Receipt of treatment with a 4-factor PCC for INR normalization due to warfarin-associated major hemorrhage

Exclusion Criteria:

* Patients treated with a PCC for an urgent invasive procedure without active hemorrhage
* Patients treated with PCC not taking a VKA
* Unavailable pre- or post-treatment INR lab values
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients administered a prothrombin complex concentrate as part of routine care for INR normalization due to a major bleed will be assessed for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Achievement of INR less than or equal to 1.5 | 60 minutes
  The number of patients achieving a goal INR of less than or equal to 1.5 within 60 minutes following administration of 4-factor fixed-dose aPCC (FEIBA VH) versus variable-dose inactivated PCC (Kcentra) for reversal of warfarin-associated major hemorrhage.

SECONDARY OUTCOMES:
Incidence of mortality or thrombotic events | 30 days
  Incidence of mortality, deep vein thrombosis, pulmonary embolism, myocardial infarction, and ischemic cerebrovascular events within 30 days following administration of 4-factor fixed-dose aPCC (FEIBA VH) or variable-dose inactivated PCC (Kcentra) for reversal of warfarin-associated major hemorrhage.

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Peksa, PharmD, Principal Investigator — Rush University Medical Center; Robert Mokszycki, PharmD, Principal Investigator — advocate christ medical center

REFERENCES:
- [Background] Junagade P, Grace R, Gover P. Fixed dose prothrombin complex concentrate for the reversal of oral anticoagulation therapy. Hematology. 2007 Oct;12(5):439-40. doi: 10.1080/10245330701448529. PMID 17852462
- [Background] Wojcik C, Schymik ML, Cure EG. Activated prothrombin complex concentrate factor VIII inhibitor bypassing activity (FEIBA) for the reversal of warfarin-induced coagulopathy. Int J Emerg Med. 2009 Nov 26;2(4):217-25. doi: 10.1007/s12245-009-0125-8. PMID 20436891
- [Background] Khorsand N, Veeger NJ, van Hest RM, Ypma PF, Heidt J, Meijer K. An observational, prospective, two-cohort comparison of a fixed versus variable dosing strategy of prothrombin complex concentrate to counteract vitamin K antagonists in 240 bleeding emergencies. Haematologica. 2012 Oct;97(10):1501-6. doi: 10.3324/haematol.2012.063701. Epub 2012 Apr 4. PMID 22491734
- [Background] Stewart WS, Pettit H. Experiences with an activated 4-factor prothrombin complex concentrate (FEIBA) for reversal of warfarin-related bleeding. Am J Emerg Med. 2013 Aug;31(8):1251-4. doi: 10.1016/j.ajem.2013.05.008. Epub 2013 Jun 10. PMID 23763937
- [Background] Sarode R, Milling TJ Jr, Refaai MA, Mangione A, Schneider A, Durn BL, Goldstein JN. Efficacy and safety of a 4-factor prothrombin complex concentrate in patients on vitamin K antagonists presenting with major bleeding: a randomized, plasma-controlled, phase IIIb study. Circulation. 2013 Sep 10;128(11):1234-43. doi: 10.1161/CIRCULATIONAHA.113.002283. Epub 2013 Aug 9. PMID 23935011